CLINICAL TRIAL: NCT02023008
Title: Convenient and Live Movement (CALM): Feasibility of Interactive Gentle Yoga for Women With Breast Cancer
Brief Title: Interactive Gentle Yoga in Improving Quality of Life in Patients With Stage I-III Breast Cancer Undergoing Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is not feasible
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00026310; NCI-2013-02387 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 01513 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Anxiety Disorder; Depression; Ductal Breast Carcinoma in Situ; Fatigue; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Anxiety Disorders; Depression; Carcinoma, Intraductal, Noninfiltrating; Fatigue; Breast Neoplasms | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (internet-based integral yoga intervention) (Experimental): Participants undergo 12 sessions of cancer-adapted integral yoga classes using an internet-based videoconferencing platform. Integral yoga includes postures, deep relaxation, breathing practices and meditation to create a profound experience of peace and well-being. Participants take part in study classes from home (or other location that is convenient for the participant and that allows them to access the internet-based classes) with two-way interaction with group instructors and members alike over 75 minutes twice weekly for 6 weeks during radiation therapy. Participants are encouraged to complete additional yoga practice sessions outside of the twice weekly study sessions.
  Interventions: Procedure: yoga therapy; Other: internet-based intervention; Other: questionnaire administration

INTERVENTIONS:
Procedure: yoga therapy — Undergo integral yoga intervention with videoconferencing
  Other Names: yoga
Other: internet-based intervention — Undergo integral yoga intervention with videoconferencing
Other: questionnaire administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies interactive gentle yoga in improving quality of life in patients with stage I-III breast cancer undergoing radiation therapy. Interactive gentle yoga may improve the quality of life in patients with breast cancer undergoing radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of implementing a 6-week biweekly yoga intervention delivered by multi-point videoconferencing in breast cancer patients undergoing radiation therapy.

SECONDARY OBJECTIVES:

I. To obtain preliminary data on changes in depression, anxiety, fatigue, sleep quality pre- and post-intervention in women with breast cancer undergoing radiation therapy.

II. To obtain preliminary data on acute effects of the yoga classes on fatigue and distress.

OUTLINE:

Participants undergo 12 sessions of cancer-adapted integral yoga classes using an internet-based videoconferencing platform. Integral yoga includes postures, deep relaxation, breathing practices and meditation to create a profound experience of peace and well-being. Participants take part in study classes from home (or other location that is convenient for the participant and that allows them to access the internet-based classes) with two-way interaction with group instructors and members alike over 75 minutes twice weekly for 6 weeks during radiation therapy. Participants are encouraged to complete additional yoga practice sessions outside of the twice weekly study sessions.

After completion of study, participants are followed up at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be newly diagnosed with a histologically or cytologically confirmed breast cancer stage I-III (ductal carcinoma in situ [DCIS] is allowed)
* Participants must have a score >= 8 on the depression subscale of the Hospital Anxiety and Depression Scale [HADS], indicating clinically significant depressive symptoms
* Participants must be:

  * >= 2 weeks post-surgery for women who have had a lumpectomy, a lumpectomy with an axillary node dissection or a mastectomy without reconstruction OR
  * >= 4 weeks post-surgery for women who have had mastectomy with reconstruction
* Participants must be scheduled to begin the standard 6-week course of radiation therapy (RT) within 4 weeks
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* For the duration of RT, participants must have access to an existing broadband internet connection and a computer (laptop or desktop; tablets are not sufficient) with a full-sized computer screen and the following specifications:

  * Windows® 8, RT, 7 Vista, XP or 2003 Server or Mac operating system (OS)® X 10.6 (Snow Leopard®) or newer
  * Internet Explorer ® 7.0 or newer, Firefox® 4.0 or newer, Safari 3.0 or newer or Chrome or newer (available for free download)
* Participants must be able to understand written/spoken English since the yoga classes will be taught in English
* Ability to understand and the willingness to sign an institutional review board (IRB)-approved written informed consent document

Exclusion Criteria:

* Participants who have practiced yoga regularly (defined as at least once per week on average) in the past 3 months
* Participants who have regularly (defined as 4 or more days per week) engaged in vigorous physical activity (i.e., causes heavy breathing, sweating, rapid fatigue; can be sustained for short periods, like running or swimming strongly) over the past 4 weeks
* Participants who are being treated with a shortened course of radiation therapy (i.e. "Canadian" fractionation less than 5 weeks, partial breast radiation therapy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Recruitment rates, calculated as the number of women enrolled divided by the number of women who screened eligible for the study | Up to week 7
Retention rates, calculated as the proportion of enrolled women who complete all study measures at each time point | Up to week 7
Adherence, measured by the total number of yoga classes attended by each participant | Up to week 7
Participants' acceptability of the intervention, including ratings of ease/difficulty of use of the videoconferencing and participating in group classes from home using the device | Up to week 7
  The proportions and 95% confidence intervals will be calculated. Descriptive statistics will be computed.
Feedback regarding the participants' experience in the study | Up to week 7
  Qualitative analysis of open-ended feedback on strengths and weaknesses of the yoga intervention and teacher, use of the multi-point videoconferencing device will be performed.

SECONDARY OUTCOMES:
Change in depression as measured by HADS | Baseline up to 7 weeks
  Computed using a mixed model analysis to account for the repeated measures on each subject.
Change in anxiety as measured by HADS | Baseline up to 7 weeks
  Computed using a mixed model analysis to account for the repeated measures on each subject.
Change in fatigue as measured by visual analogue scale and Functional Assessment of Cancer Therapy-Fatigue | Baseline up to 7 weeks
  Computed using a mixed model analysis to account for the repeated measures on each subject. Assessed by calculating the difference in the post and pre scores for each session, and then examining whether there is a time effect using a mixed model.
Change in sleep quality as measured by Pittsburgh Sleep Quality Inventory | Baseline up to 7 weeks
  Computed using a mixed model analysis to account for the repeated measures on each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Danhauer, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States